CLINICAL TRIAL: NCT03722602
Title: Effect of Rehabilitation on the Body Composition in Patients With Stroke
Brief Title: Body Composition of People After a Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rzeszow (Other)
Responsible Party: Principal Investigator, Justyna Leszczak, Principal Investigator, University of Rzeszow
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Stroke-BodyComposition
Record Dates: First submitted 2018-05-22; First posted 2018-10-29 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Rehabilitation; Stroke; Body Composition
Keywords: stroke; BMI; body composition; functional scales
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rehabilitation group (Experimental): Patients with stroke receiving standard inpatient rehabilitation for five weeks
  Interventions: Other: Standard rehabilitation after stroke

INTERVENTIONS:
Other: Standard rehabilitation after stroke — The program of the rehabilitation was designed specifically for each patient. It was prepared to match the patient's functional status and the defined goals. The subjects participated in exercise five days per week, for five weeks. During their stay at the Clinic, the patients took part in morning exercise and received individual practice, based on neuro-developmental treatment (Bobath concept), and proprioceptive neuromuscular facilitation (PNF) method, addressing the impaired motor abilities; if it was needed they also performed exercise based on equipment using biological feedback: Balance Trainer (static and dynamic parapodium) and Pablo system designed for upper limb training.

SUMMARY:
The study enabled assessment of changes in body mass composition, metabolic syndrome and lipid profile in patients after stroke, following rehabilitation in hospital.

DETAILED DESCRIPTION:
Stroke is estimated to affect 24-54% of the global population and is one of the leading causes of death. According to World Health Organization over one billion people worldwide are overweight, and approximately 300 million people are obese. The main factors contributing to this situation include insufficient physical activity and unhealthy diet. Among the major consequences of obesity in adults one can distinguish metabolic syndrome and cardiovascular diseases.

Therefore, measurements were performed to identify changes in body mass composition (body fat, visceral fat level, muscle mass, total body water, metabolic syndrome, lipid profile) in subjects after stroke following rehabilitation at hospital.

The study was carried at the Clinical Rehabilitation Ward with Early Neurological Rehabilitation Unit, at the Clinical Hospital in Rzeszów, Poland. The measurements were performed from June 2015 to March 2017. During that time the total of 1,143 patients received treatment and rehabilitation at the clinic. These included 403 patients after stroke. The subjects were examined three times. In accordance with inclusion and exclusion criteria 128 subjects were qualified for the first exam. The second exam took into account 114 subjects and finally 100 patients with stroke participated in the third exam. The analyses took into account the data obtained from the 100 subjects who took part in all the exams. Body mass composition was assessed in all the subjects with Tanita MC 780 MA analyzer, whose operation is based on Bioelectrical impedance analysis (BIA). The subjects' height was measured with the stadiometer PORTSTAND 210. Rehabilitation outcome was assessed with Barthel index, Berg scale, Ashworth scale, Brunnström scale, Rankin scale and symmetry index for lower limb weight distribution (Ws).

In addition, waist and hip circumference were measured and WHR was calculated. The above parameters were assessed three times:

Exam I took place upon admission to hospital Exam II on the day the patient was discharged from hospital Exam III was performed 12 weeks after discharge from hospital during a follow-up visit.

The follow-up visit, 12 weeks after discharge from hospital, was meant to determine whether the effects of rehabilitation persisted for 12 weeks after discharge from hospital.

Other parameters examined included: LDL, HDL, total cholesterol, TG, atherogenic index, CRP, and serum glucose level. Blood for the tests was drawn from basilic vein by medical personnel at the Rehabilitation Clinic. The test was performed twice: upon admission to the Clinic and following 5-week rehabilitation at the hospital.

ELIGIBILITY:
Inclusion criteria:

* Stroke experienced.
* Ability to stand without assistance.
* Ability to walk without aid.
* No impairments in higher mental functions
* Patient's informed, voluntary consent to participate in the study.

Exclusion criteria:

* Lack of patient's consent to participate in the study
* Lack of ability to stand without assistance.
* Ischemic lesion located in the cerebellum and brain stem.
* Metal, electronic implants.
* Epilepsy.
* Pregnancy.
* Menstruation, in females.
* Limb injuries incurred following stroke onset, prior to the exam.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Change Body composition assessment (fat mass, visceral fat level , muscle tissue, fat free mass , water content in the body) subjected to bioelectrical impedancy analysis - Tanita 780. | at baseline, immediately after treatment completion, and 12 weeks after treatment completion
  Assessment of body composition (bioelectrical impedancy analysis - Tanita 780) Change from Baseline body composition at 5 weeks between baseline, after the end of protocol treatment, and 12 weeks after the end of the protocol treatment.

SECONDARY OUTCOMES:
Assessment of functional status was assessed using the Barthel Index. The subjects could score the maximum of 100 points. | at baseline, immediately after treatment completion, and 12 weeks after treatment completion
  Activities of daily living were assessed using Barthel Index. The subjects could score the maximum of 100 points.
  A maximum of 100 points can be obtained on the Barthel scale. There are three assessment ranges: getting from 0 to 20 points. means total dependence, from 20 to 80 points. means that to some extent the patient needs help from others, and the assessment in the border is 80 to 100 points. means that with a little help the patient can function alone.
  0-20 points patient's condition "light" 21-85 points - "medium-heavy" patient condition 86-100 points - patient condition "very heavy"
Balance was assessed using Berg Balance Scale (BBS) | at baseline, immediately after treatment completion, and 12 weeks after treatment completion
  Balance was assessed using Berg balance scale (BBS)
  Berg Balance Scale
  Description:
  14-item scale designed to measure balance
  (1. Sitting to standing 2. Standing unsupported 3. Sitting unsupported 4. Standing to sitting 5. Transfers 6. Standing with eyes closed 7. Standing with feet together 8. Reaching forward with outstretched arm 9. Retrieving object from floor 10. Turning to look behind 11. Turning 360 degrees 12. Placing alternate foot on stool 13. Standing with one foot in front 14. Standing on one foot)
  Scoring: A five-point ordinal scale, ranging from 0-4. "0" indicates the lowest level of function and "4" the highest level of function. Score the LOWEST performance. Total Score = 56
  Interpretation: 41-56 = independent 21-40 = walking with assistance 0 -20 = wheelchair bound
Assessment of muscle tone (spasticity) was examined with modified Ashworth scale. | at baseline, immediately after treatment completion, and 12 weeks after treatment completion
  Increased muscle tone (spasticity) was examined with modified Ashworth scale. This is a six-point scale modified to include grade 1.
  0: No increase in muscle tone
  1. Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension 1+: Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM
  2. More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved
  3. Considerable increase in muscle tone, passive movement difficult
  4. Affected part(s) rigid in flexion or extension
Assessment of paretic limb function was assessed using the Brunnström scale. | at baseline, immediately after treatment completion, and 12 weeks after treatment completion
  Motor performance (function) of extremities was assessed using Brunnström scale. This is a six-point scale designed to assess performance (function) of paretic extremities
Assessment of symmetry index for lower limb weight distribution | at baseline, immediately after treatment completion, and 12 weeks after treatment completion
  Symmetry index for lower limb weight distribution (Ws) was calculated based on data obtained in tandem balance test, where the higher value was divided by the lower value. Normal index value, which was assumed in the range from 1.00 to 1.15, reflects the fact that weight is evenly distributed between legs, with permissible deviation up to 4-5 kilograms
Assessment of disability level, using the modified Rankin scale (MRS) | at baseline, immediately after treatment completion, and 12 weeks after treatment completion
  Assessment of disability using the modified Rankin scale (MRS)
  Score Description 0 - No symptoms at all
  1- No significant disability despite symptoms; able to carry out all usual duties and activities 2 - Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance 3 - Moderate disability; requiring some help, but able to walk without assistance 4 - Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance 5 - Severe disability; bedridden, incontinent and requiring constant nursing care and attention 6 - Dead TOTAL (0-6): _______
Changes in blood parameter: HDL | at 5 weeks between baseline, after the end of protocol treatment,
  Blood for the tests was drawn from basilic vein by medical personnel at the Rehabilitation Clinic.
  HDL level:
  Men:
  Less than 35 mg / dL (0.9 mmol / L) high risk of heart disease.
  Women:
  Lower than 45 mg / dL (1.2 mmol / L) high risk of heart disease. 60 mg / dL (1.56 mmol / L) and above. High HDL cholesterol.
Changes in blood parameter: LDL | at 5 weeks between baseline, after the end of protocol treatment
  Blood for the tests was drawn from basilic vein by medical personnel at the Rehabilitation Clinic.
  LDL level:
  Less than 100 mg / dL (2.6 mmol / L) Norm 100 - 129 mg / dL (2.63.34 mmol / L) Above the norm 130 - 159 mg / dL (3.36 - 4.13 mmol / L) Limit 160 - 189 mg / dL (4.14 - 4.90 mmol / L) High 190 mg / dL (4.91 mmol / L) and above Very high
Changes in blood parameter: total cholesterol | at 5 weeks between baseline, after the end of protocol treatment
  Blood for the tests was drawn from basilic vein by medical personnel at the Rehabilitation Clinic.
  Total Cholesterol level:
  Less than 200 mg / dL (5.17 mmol / L) Norm 200 - 239 mg / dL (5.17 - 6.18 mmol / L) Elevated level 240 mg / dL (6.21 mmol / L) High risk of heart disease
Assessment of WHR | at 5 weeks between baseline, after the end of protocol treatment, and 12 weeks after treatment completion
  The type of obesity is assessed with the so-called waist-to-hip ratio (WHR), which shows the proportion of waist circumference and hip circumference. WHR specifies the location of excessive fat and makes it possible to identify two main types of obesity: visceral obesity (characteristic for men), connected with accumulation of fat in the abdominal cavity and upper part of the body, and gynoid obesity (gluteal-femoral), more common in women.
Assessment of metabolic syndrome | at 5 weeks between baseline, after the end of protocol treatment
  Metabolic syndrome (polymetabolic syndrome, syndrome X, insulin resistance syndrome, Reaven syndrome) - a set of interrelated factors significantly increasing the risk of atherosclerosis and type 2 diabetes, as well as their vascular complications.
  Abdominal (central) obesity
  At least three of the following five abnormalities must be identified to formulate a diagnosis:
  abdominal obesity (waist circumference in men from Europe ≥ 94 cm, and in women ≥ 80 cm) and additionally co-existing two of the following abnormalities: triglycerides ≥ 150 mg/dl or dyslipidaemia related treatment cholesterol HDL < 40 mg/dl in males < 50 mg/dl in females or dyslipidaemia related treatment arterial pressure ≥ 130/85 mm Hg or arterial pressure related treatment fasting glycaemia ≥ 100 mg/dl or type 2 diabetes treatment
Changes in blood parameter: TG | at 5 weeks between baseline, after the end of protocol treatment,
  Blood for the tests was drawn from basilic vein by medical personnel at the Rehabilitation Clinic.
  TG level:
  Below 150mg / dL (1.69mmol / L) Norm 150 - 199 mg / dL (1.69 - 2.25 mmol / L) Limit 200 - 499 mg / dL (2.26 - 5.63 mmol / L) High Above 500 mg / dL (5.64 mmol / L) Very high
Changes in blood parameter: atherogenic index | at 5 weeks between baseline, after the end of protocol treatment,
  Blood for the tests was drawn from basilic vein by medical personnel at the Rehabilitation Clinic.
  atherogenic index level
  * in men below 4.5 (below 3.5 after myocardial infarction)
  * in women below 4.0 (below 3.0 after myocardial infarction)
Changes in blood parameter: CRP | at 5 weeks between baseline, after the end of protocol treatment,
  Blood for the tests was drawn from basilic vein by medical personnel at the Rehabilitation Clinic.
  CRP level:
  * CRP below 5 mg / l (up to 10 mg / l - in obese people with hypertension) norm
  * CRP above 40 mg / l - may indicate a mild viral infection or pregnancy;
  * CRP above 200 mg / l - bacterial inflammation develops in the body;
  * CRP above 500 mg / l - takes place in the situation of very serious infections with basic and bacterial infections and burns.
Changes in blood parameter: serum glucose | at 5 weeks between baseline, after the end of protocol treatment,
  Blood for the tests was drawn from basilic vein by medical personnel at the Rehabilitation Clinic.
  serum glucose level: From 70 to 99 mg / dL (from 3.9 to 5.5 mmol / L) Normal glucose level From 100 to 125 mg / dL (from 5.6 to 6.9 mmol / L) Abnormal fasting glucose (pre-diabetes) From 126 mg / dL (7.0 mmol / L) Diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Justyna Leszczak, PhD, Principal Investigator — University of Rzeszow
Locations (1):
- University of Rzeszów, Rzeszów, Poland